CLINICAL TRIAL: NCT00413101
Title: An Open-Label Study to Investigate Improvement in Heart Function After Complete Anemia Correction With NeoRecormon in Patients With End-Stage Renal Disease Already Receiving Sub-Optimal Doses of NeoRecormon
Brief Title: A Study of NeoRecormon (Epoetin Beta) in Patients With End Stage Renal Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20201
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: epoetin beta [NeoRecormon]

INTERVENTIONS:
Drug: epoetin beta [NeoRecormon] — At a dose to achieve and maintain an Hb level of 120-135g/L

SUMMARY:
This single arm study will determine the effects of complete anemia correction in anemic patients with end-stage renal disease currently receiving suboptimal doses of NeoRecormon. Patients on dialysis receiving NeoRecormon, and with a hemoglobin level <105g/L, will be treated with subcutaneous NeoRecormon at a dose determined by the investigator in order to reach (within 3 months) and maintain a hemoglobin level in the range of 120-135g/L. Heart function and quality of life will be measured before and after anemia correction. The anticipated time on study treatment is 3-12 months, and the target sample size is 100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* end-stage renal disease;
* on renal dialysis >= 3 months;
* receiving NeoRecormon treatment >= 3 months;
* Hb stable and <105g/L, and LVMI >160g/m2.

Exclusion Criteria:

* unstable hypertension, myocardial infarction, unstable angina pectoris or risk of deep vein thrombosis in last 6 months;
* use of any ESA other than NeoRecormon;
* acute infection;
* use of iv NeoRecormon.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Hb level, BP. | Throughout study
LVMI ejection fraction, ejection fraction. | 12 months

SECONDARY OUTCOMES:
SAEs, AEs leading to withdrawal, AEs related to NeoRecormon. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Novi Sad, Serbia